CLINICAL TRIAL: NCT00907335
Title: A Multi-Center, Double Blind, Vehicle Controlled, Study of Retin-A Micro 0.04% in the Treatment of Pediatric Acne Vulgaris in Children, Ages 9 to 11 Years of Age
Brief Title: A Study of Acne Treatment in Children Ages 9 to 11
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA-P-6397
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Results first posted 2011-03-11 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Acne Vulgaris
Keywords: acne; irritation; objective sensory methods
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Retin-A Micro (Experimental): Retin-A Micro 0.04% facial acne treatment used once daily
  Interventions: Drug: Retin-A Micro 0.04% facial acne treatment
- Vehicle Control (Placebo Comparator): Color matched facial gel vehicle control used once daily
  Interventions: Drug: Vehicle control

INTERVENTIONS:
Drug: Retin-A Micro 0.04% facial acne treatment — Retin-A Micro 0.04% facial acne treatment used once daily
  Other Names: facial acne treatment
  Arms: Retin-A Micro
Drug: Vehicle control — Color-matched facial gel vehicle control used once daily
  Other Names: placebo
  Arms: Vehicle Control

SUMMARY:
A study to determine if using Retin-A Micro 0.04% as facial acne treatment in patients ages 9 to 11 is safe and efficacious.

DETAILED DESCRIPTION:
Approximately 100 female and male subjects, aged from 9 to 11 years of age, will be enrolled in this randomized, double blind, multi-center study.

Following satisfaction of entry criteria and screening procedures, subjects will receive either RETIN-A MICRO 0.04% or a color matched gel vehicle for once daily use during the 12-week treatment period. Subjects will be monitored for safety throughout the study and for signs and symptoms of local irritation at baseline, and at weeks 2, 4, 6, 8, 10 and again at study completion, week 12.

Efficacy will be assessed by facial lesion counts and by utilizing scales for Investigator's Global Evaluation of Acne Severity (IGA #1 and IGA #2) and Investigator's Global Assessment of Improvement (IGA #3). All efficacy parameters with the exception of IGA #3 will be measured at baseline and weeks 2, 4, 6, 8, 10 and 12. The Investigator's Global Assessment of Improvement (IGA #3) will be done at Week 12 only. At selected sites, photographs will be taken at Baseline and weeks 2, 4, 8 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-nursing females, 9 to 11 years, with facial pediatric acne vulgaris
* Minimum of 20 non-inflammatory lesions (open and closed comedones)
* Minimum of 30 total facial lesions (sum of inflammatory and non-inflammatory)
* Must have at least a rating of grade 3 on the Investigator Global Assessment Scale for acne severity (IGA #1) at baseline

Exclusion Criteria:

* Known sensitivity to any of the ingredients in the study medication;
* Any nodulocystic acne lesions
* Use of acne devices or systemic therapy with antibiotics within two months prior to start and throughout the duration of the study
* Use of systemic therapy with retinoids within four months prior to study start and throughout the duration of the study
* Topical use of topical retinoids within two weeks prior to study start and throughout the duration of the study
* Topical use of antibiotics, steroids and/or other non-retinoid topical acne products within two weeks prior to study start and throughout the duration of the study
* Use of an experimental drug or device within 60 days prior to study start;
* Use of hormonal therapy within 3 months prior to study start
* History of evidence of other skin conditions or diseases that may require concurrent therapy or may interfere with the evaluation of the study medication
* Any significant medical conditions that could confound the interpretation of the study
* History of/or current facial skin cancer
* Inability to refrain from use of all facial products other than those supplied by the study, while participating in the study
* No use of tanning booths, sun lamps, etc.
* Subject is a family member of the employee or the investigator

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rossi, MD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (12):
- United States (12):
  - Encino Research Center, Encino, California
  - Children's Hospital and Health Center, San Diego, California
  - Department of Dermatology, University of Miami, Miami, Florida
  - Department of Dermatology, Northwestern University, Chicago, Illinois
  - Dermatology Associates, Louisville, Kentucky
  - UMDNJ-RWJ Medical School, Somerset, New Jersey
  - SUNY Downstate Medical Center Department of Dermatology, Brooklyn, New York
  - Dermatology Research Associates, Cincinnatti, Ohio
  - Skin Study Center, Broomall, Pennsylvania
  - Yardley Dermatology Associates, Yardley, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - University of Texas Medical School at Houston, Houston, Texas

REFERENCES:
- [Derived] Eichenfield LF, Hebert AA, Schachner L, Paller AS, Rossi AB, Lucky AW. Tretinoin microsphere gel 0.04% pump for treating acne vulgaris in preadolescents: a randomized, controlled study. Pediatr Dermatol. 2012 Sep-Oct;29(5):598-604. doi: 10.1111/j.1525-1470.2012.01811.x. Epub 2012 Jun 19. PMID 22712470
- See also: FDA's Drug Finder — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Retin-A Micro | Vehicle Control
Started | 55 | 55
Completed | 47 | 54
Not Completed | 8 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 4 | 1
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retin-A Micro | Vehicle Control | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Customized [Number; unit: participants]
  9 years | 5 | 4 | 9
  10 Years | 21 | 17 | 38
  11 Years | 29 | 34 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 38 | 82
  Male | 11 | 17 | 28
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110
Subject Reached Puberty [Number; unit: Participants]
  Yes | 17 | 21 | 38
  No | 38 | 34 | 72
Fitzpatrick Score [Number; unit: Participants] — Skin type is categorized according to the Fitzpatrick skin type scale, which ranges from very fair (skin type I) to very dark (skin type VI).
  Participants
    I | 2 | 1 | 3
    II | 17 | 12 | 29
    III | 11 | 16 | 27
    IV | 14 | 15 | 29
    V | 8 | 9 | 17
    VI | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Non-inflammatory Lesion Count
Description: Change from Baseline to Week 12 (Week 12 minus Baseline) in the total non-inflammatory acne lesion count. Facial acne lesion counts consisted of non-inflammatory lesions and inflammatory lesions. The total non-inflammatory acne lesion count is the sum of open and closed comedones, change from Baseline was calculated as the value after Baseline minus the baseline value, and negative changes indicated lesion improvement.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Retin-A Micro | Vehicle Control
Number analyzed (Participants) | 47 | 54
Lesions | -19.9 (4.13) | -9.7 (4.42)

2. Secondary Outcome: Change From Baseline in Lesion Counts
Description: Change from baseline in Lesion Count by the following categories: Facial acne lesion counts consisted of non-inflammatory lesions and inflammatory lesions. Inflammatory lesions were the sum of papules and pustules. Total lesions were the sum of non-inflammatory and inflammatory lesions, plus nodules/cysts. For each lesion type, change from Baseline was calculated as the value after Baseline minus the baseline value, and negative changes indicated lesion improvement.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Retin-A Micro | Vehicle Control
Number analyzed (Participants) | 47 | 54
Lesions
  Comedones | -19.85 (4.13) | -9.67 (4.42)
  Inflammatory | -0.63 (1.16) | 0.54 (1.23)
  Total Lesions | -21.87 (4.64) | -10.88 (4.97)
  Open Comedones | -4.10 (1.77) | -2.86 (1.87)
  Closed Comedones | -15.16 (2.92) | -6.09 (3.14)
  Papules | -0.62 (0.75) | -0.48 (0.79)
  Pustules | -0.17 (0.77) | 1.04 (0.81)

3. Secondary Outcome: Measurement of Success 1
Description: Participants achieving success according to the Investigator Global Assessment (IGA #1) - (Pediatric Acne Scale) has ordinal response categories identified as clear (0), almost clear (1), mild (2), moderate (3), severe (4), and very severe (5). The number of participants for which treatment was considered successful was based on 2 criteria: 1) improvement by at least 2 grades from the baseline score, and 2) ratings of clear or almost clear.
Time Frame: Week 12
Measure: Number; unit: Participants
Arm/Group | Retin-A Micro | Vehicle Control
Number analyzed (Participants) | 47 | 54
Participants
  Clear/Almost Clear | 11 | 11
  At Least 2 Grades Improvement | 15 | 12

4. Secondary Outcome: Measurement of Success 2
Description: Participants achieving success according to dichotomized Investigator Global Assessment (IGA) scores - Food and Drug Administration Score (IGA#2) The IGA #2 (static 5 point scale recommended in the FDA acne guidelines) has ordinal response categories identified as clear (0), almost clear (1), mild (2), moderate (3), and severe (4). The number of participants for which treatment was considered successful was based on 2 criteria: 1) improvement by at least 2 grades from the baseline score, and 2) ratings of clear or almost clear.
Time Frame: Week 12
Measure: Number; unit: Participants
Arm/Group | Retin-A Micro | Vehicle Control
Number analyzed (Participants) | 47 | 54
Participants
  Clear/Almost Clear | 10 | 10
  At Least 2 Grades Improvement | 8 | 8

5. Secondary Outcome: Measurement of Success 3
Description: Participants achieving success according to Investigator Global Assessment (IGA#3) scores. At Week 12, the IGA #3 rated the subject's improvement over Baseline by using the following categories: Excellent, Good, Fair, No Change, Worse. The number of participants for which treatment was considered successful was based on the IGA #3 success criteria defined as achievement of "Excellent" or "Good" scores.
Time Frame: Week 12
Measure: Number; unit: Participants
Arm/Group | Retin-A Micro | Vehicle Control
Number analyzed (Participants) | 47 | 54
Participants
  Success | 31 | 27
  No Success | 16 | 27

6. Secondary Outcome: Global Assessment
Description: Participants showing improvement from baseline in the Investigator's Global Assessment, in the Intent to Treat population using the Last Available Measurement and imputation technique of Last Observation Carried Forward, rating the subject's improvement over Baseline by using the following categories: Excellent, Good, Fair, No Change, Worse.
Time Frame: Baseline to Week 12
Measure: Number; unit: Participants
Arm/Group | Retin-A Micro | Vehicle Control
Number analyzed (Participants) | 47 | 54
Participants
  Excellent | 12 | 7
  Good | 19 | 20
  Fair | 11 | 9
  No Change | 5 | 18
  Worse | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: Subjects asked if they experienced adverse events at each visit.
Arm/Group | Retin-A Micro | Vehicle Control
Serious Adverse Events (participants affected / at risk) | 0/55 | 1/55
Other Adverse Events (participants affected / at risk) | 25/55 | 7/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retin-A Micro (N=55) | Vehicle Control (N=55)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retin-A Micro (N=55) | Vehicle Control (N=55)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3)
Pharyngitis Streptococcal (Infections and infestations) | 3 (3) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 3 (3)
Sunburn (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 13 (13) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less